CLINICAL TRIAL: NCT05857592
Title: Adapting Self-report Instruments for People With Intellectual Disability to Improve Cognitive Accessibility - Putting Guidelines to the Test
Brief Title: Improving the Cognitive Accessibility of Self-reports for People With ID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koraal (Other)
Collaborators: University of Amsterdam (Other); Zuyd University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Roel Kooijmans, Senior Researcher, Koraal
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Koraal-ABAS-Kooijmans
Record Dates: First submitted 2023-03-15; First posted 2023-05-12 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Mild Intellectual Disability; Borderline Intellectual Functioning
Keywords: self-report questionnaires; inclusive diagnostics; easy-read language; adaptive functioning

STUDY DESIGN:
Intervention Model Description: A mixed-method repeated-measures design will be used: data are collected using both qualitative and quantitative methods at two points in time (before and after adaptation) from the same participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Persons with Mild Intellectual Disability (MID) or Borderline Intellectual Functioning (BIF) complete the ABAS-3 in assisted form on two occasions: the original version the first time and an adapted version after a few weeks.
  Interventions: Diagnostic Test: Adaptive functioning self-report questionnaire; Diagnostic Test: Adaptive functioning self-report questionnaire - adapted

INTERVENTIONS:
Diagnostic Test: Adaptive functioning self-report questionnaire — A self-report questionnaire for assessing level of adaptive functioning
Diagnostic Test: Adaptive functioning self-report questionnaire - adapted — A self-report questionnaire for assessing level of adaptive functioning, adapted to the communication level of the participant

SUMMARY:
In the proposed study, the investigators aim to investigate whether the existing ABAS-3 self-report questionnaire is suitable to be completed meaningfully by individuals who are perceived as having mild intellectual disability (55<IQ<85) based on cognitive impairment. Based on the participants' experiences and researchers' expertise, the investigators develop a 'more inclusive' self-report version. The investigators then look at the extent to which participants indicate that they understand this version better, based on user experiences and limited psychometric research. In doing so, the investigators also compare the outcomes of the self-report and informant-report variant.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Last known Total Intelligence Quotient (TIQ) 55 - 85
* Receiving support from a care organization for persons with ID.
* A care worker who knows the participant for at least a year and knows him well enough tot complete the informant version of the ABAS-3 is available.

Exclusion Criteria:

• Severe physical or sensory impairment limiting ability to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Scoring comprehension - T0 | At baseline (T0)
  Degree to which the qualitative information provided by the participant aligns with the self-reported score on the original version of the ABAS-3 (Adaptive Behaviour Assessment System - Third Edition) questionnaire. Outcomes are 0, scores align, -1, scores are lower than answer would suggest, +1, score is higher than answer would suggest.
Scoring comprehension - T1 | Approximately 8 weeks after baseline (T1)
  Degree to which the qualitative information provided by the participant aligns with the self-reported score on the original version of the ABAS-3 (Adaptive Behaviour Assessment System - Third Edition) questionnaire. Outcomes are 0, scores align, -1, scores are lower than answer would suggest, +1, score is higher than answer would suggest.
Text comprehension - cognitive interviews T0 | At baseline (T0)
  Level of verbal understanding of questions in the questionnaire - qualitative analysis of answers from cognitive interviews during assessment of the ABAS-3 (Adaptive Behaviour Assessment System - Third Edition). Terms and concepts that were misinterpreted, participant utterings of confusion of statements of difficulty
Text comprehension - cognitive interviews T1 | Approximately 8 weeks after baseline (T1)
  Level of verbal understanding of questions in the questionnaire - qualitative analysis of answers from cognitive interviews during assessment of an adapted version of the ABAS-3 (Adaptive Behaviour Assessment System - Third Edition). Terms and concepts that were misinterpreted, participant utterings of confusion of statements of difficulty.
Comprehension of instructions - cognitive interviews T0 | At baseline (T0)
  Level of verbal understanding of the instructions in the questionnaire - original version of the ABAS-3 (Adaptive Behaviour Assessment System - Third Edition). Number of elements that were correctly identiefied (out of possible 10).
Comprehension of instructions - cognitive interviews T1 | Approximately 8 weeks after baseline (T1)
  Level of verbal understanding of the instructions in the questionnaire - adapted version of the ABAS-3 (Adaptive Behaviour Assessment System - Third Edition). Number of elements that were correctly identiefied (out of possible 10).
Overall difficulty score - T0 | At baseline (T0)
  Likert scale rating of the overall difficulty of items of original version of the ABAS-3 (Adaptive Behaviour Assessment System - Third Edition) by participants (from 1. very easy - 5. very difficult)
Overall difficulty score - T1 | Approximately 8 weeks after baseline (T1)
  Likert scale rating of the overall difficulty of items of adapted version of the ABAS-3 (Adaptive Behaviour Assessment System - Third Edition) by participants (from 1. very easy - 5. very difficult)

SECONDARY OUTCOMES:
Self-reported Adaptive Functioning - original ABAS-3 scores | At baseline (T0)
  The ABAS-3 (Adaptive Behaviour Assessment System - Third Edition) is an observational scale that measures adaptive behaviour. Both self-report and informant report versions are available. In the context of the current study, a 30-item abbreviated version is used. Composite scores are calculated: a total score and three domain scores (conceptual, social and practical domain). Scores range from 0-90 for the total scale and 0-30 for each domain scale. Higher scores indicate better adaptive functioning.
Self-reported Adaptive Functioning - adapted ABAS-3 scores | Approximately 8 weeks after baseline (T1)
  The ABAS-3 (Adaptive Behaviour Assessment System - Third Edition) is an observational scale that measures adaptive behaviour. Both self-report and informant report versions are available. In the context of the current study, a 30-item abbreviated version is used. Composite scores are calculated: a total score and three domain scores (conceptual, social and practical domain). Scores range from 0-90 for the total scale and 0-30 for each domain scale. Higher scores indicate better adaptive functioning.
  The second time participants complete the ABAS (approximately 8 weeks after baseline, T1), an adapted version is used, with language and design adapted to the comprehension level of participants according to the outcomes at baseline (T0).
Informant-reported Adaptive Functioning - original ABAS-3 scores | At baseline (T0)
  The ABAS-3 (Adaptive Behaviour Assessment System - Third Edition) is an observational scale that measures adaptive behaviour. Both self-report and informant report versions are available. In the context of the current study, a 30-item abbreviated version is used. Composite scores are calculated: a total score and three domain scores (conceptual, social and practical domain). Scores range from 0-90 for the total scale and 0-30 for each domain scale. Higher scores indicate better adaptive functioning.
  For the informant-report an adapted version of the original is used; the adaptations for the self-report version are replicated for the informant version.
Informant-reported Adaptive Functioning - adapted ABAS-3 scores | Approximately 8 weeks after baseline (T1)
  The ABAS-3 (Adaptive Behaviour Assessment System - Third Edition) is an observational scale that measures adaptive behaviour. Both self-report and informant report versions are available. In the context of the current study, a 30-item abbreviated version is used. Composite scores are calculated: a total score and three domain scores (conceptual, social and practical domain). Scores range from 0-90 for the total scale and 0-30 for each domain scale. Higher scores indicate better adaptive functioning.
  For the informant-report an adapted version of the original is used; the adaptations for the self-report version are replicated for the informant version.
Self-reported Adaptive functioning - SCAF | At baseline (T0)
  The SCAF (Screener for Adaptive Functioning) is a screening questionnaire for adaptive functioning for individuals who may have MID or BIF. The SCAF yields a total AF score (min 0 - max 24), with higher scores indicating better adaptive functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Roel Kooijmans, MSc, Principal Investigator — Koraal
Locations (1):
- Koraal, Sittard, L, Netherlands

IPD SHARING:
Plan to Share IPD: No
Study data are highly specific for this study and not relevant for sharing with other researchers, except for validation of results in exceptional circumstances. When required, relevant data will be made available upon request to reviewers or auditors, subject to privacy regulations. Only anonymized data will be shared.

REFERENCES:
- [Background] Kooijmans, R., Mercera, G., Langdon, P. E., & Moonen, X. (2022). The adaptation of self-report measures to the needs of people with intellectual disabilities: A systematic review. Clinical Psychology: Science and Practice.